CLINICAL TRIAL: NCT01492452
Title: Standard Guidelines Impact of Nursing Anxiety of Parents of Children Undergoing Cardiac Surgery: Randomized Clinical Trial
Brief Title: The Anxiety of Parents of Children Undergoing Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Cardiologia do Rio Grande do Sul (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single
Other Study IDs: UP4555/10
Record Dates: First submitted 2011-12-13; First posted 2011-12-15 (Estimated); Last update posted 2011-12-15 (Estimated); Status verified 2011-12

CONDITIONS: Anxiety
Keywords: guidelines for nursing; anxiety; cardiac surgery; pediatrics
MeSH Terms: conditions — Anxiety Disorders | interventions — Nursing

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- guidelines (No Intervention): 22 parents in the intervention group were randomized and received standardized guidelines for nursing:The guidelines took around an hour and involved pre-operative care such as bathing with detergent solution, pre-anesthetic administration (as prescribed), preoperative fasting (as prescribed), clothing, hygiene care and nail oral. They were also provided information on the endotracheal tube, tubes, catheters, epicardial pacemaker wires and electrodes to be used in the perioperative period and which remain for some period after surgery, as well as possible complications.
  Interventions: Other: standardized guidelines for nursing

INTERVENTIONS:
Other: standardized guidelines for nursing — Information was provided regarding the preoperative preparation of the child, the same conditions and in the postoperative period, as well as information relating to housing and food for the parents. The conventional orientation took about 15 minutes.
  Other Names: parents aged over 18 years

SUMMARY:
This is a randomized clinical trial. The population consisted of parents of children undergoing cardiac surgery from December 2010 to April 2011. We included parents aged over 18 years, and the following were considered exclusion criteria: inability to understand and/or answer the questions for any reason, parents of children undergoing surgery for insertion of the pacemaker and defibrillator, surgical death and not take up the case. 22 parents in the intervention group were randomized and received standardized guidelines for nursing and 22 parents participated in the control group received the guidelines and routine of the institution. Anxiety was assessed using the STAI State-Trait Inventory in the preoperative period and 48 hours after surgery the child.

DETAILED DESCRIPTION:
anxiety

ELIGIBILITY:
Inclusion Criteria:

* We included parents aged over 18 years

Exclusion Criteria:

* inability to understand and/or answer the questions for any reason,
* parents of children undergoing surgery for insertion of the pacemaker and defibrillator,
* surgical death and not take up the case

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2010-12; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
anxiety inventory | five months
  STAI State-Trait Inventory

CONTACTS AND LOCATIONS:
Overall Officials: M A Moraes, Phd, Principal Investigator — Institute of Cardiology